CLINICAL TRIAL: NCT03151850
Title: The Diversity of the Fungal and Bacterial in Colon Mucosa of Patients With Ulcerative Colitis Associated Different Clinical Classification
Brief Title: The Diversity of the Fungal and Bacterial in Colon Mucosa of Patients With Different Degree of Inflammation of Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiuli Zuo (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, Deputy director of the physician, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2015SDU-QILU-G004
Record Dates: First submitted 2016-12-19; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Ulcerative Colitis
Keywords: fungal; mucosa; diversity; Basidiomycete
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ulcerative colitis: We analysed the diversity of the fungal and bacterial in patients with Ulcerative Colitis (UC). We take 2 pieces of biopsies in the sigmoid colon mucosa inflammation area during the colonoscopy and then perform gene sequencing.
  Interventions: Other: ulcerative colitis
- Control: Analysing the diversity of the fungal and bacterial in patients without ulcerative colitis. We take 2 pieces of biopsies in the sigmoid colon mucosa during the colonoscopy and then perform gene sequencing.
  Interventions: Other: Control

INTERVENTIONS:
Other: ulcerative colitis — We take 2 pieces of biopsies in the sigmoid colon mucosa inflammation area during the colonoscopy and then perform gene sequencing.
  Other Names: Patients With ulcerative colitis
  Groups: ulcerative colitis
Other: Control — We take 2 pieces of biopsies in the sigmoid colon mucosa during the colonoscopy and then perform gene sequencing.
  Other Names: Patients Without ulcerative colitis
  Groups: Control

SUMMARY:
We analyzed the diversity of the fungal and bacterial within colon mucosa between patients with different degree of inflammation of Ulcerative Colitis.

DETAILED DESCRIPTION:
In recent years, the relationship of intestinal fungus with inflammatory bowel disease was gradually revealed. We divided the patients with ulcerative colitis into three groups on the basis of World Gastroenterology Organisation (WGO) classification about inflammation degree and progress classification and established the healthy control group. Analyzing the diversity of the fungal and bacterial within colon mucosa between patients with different clinical classification, for example, the proportion of bacteria and fungi, the proportion of candida albicans, the proportion of yeasts, and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients at our tertiary care medical center, aged between 18 and 80 years, scheduled to undergo surveillance colonoscopy.
* The patients with ulcerative colitis for ulcerative colitis group.
* The patients without ulcerative colitis for control group.
* 18-80 years.

Exclusion Criteria:

* Using antibiotics, glucocorticoid and immunosuppressants wintin one month.
* There are contraindications for enteroscopy and biopsy.
* There are other intestinal diseases.
* Pregnancy or breast-feeding women.
* Patients with serious lung disease and mental illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients under endoscopic surveillance or examination at Qilu Hospital were considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
fungus detection rate | 6 months
  Fungi detection rate was defined as the percentage of patients in whose colonic mucosa at least one kind of fungus were identified.
yeasts detection rate | 6 months
  Yeasts detection rate was defined as the percentage of patients in whose colonic mucosa yeasts were identified.
candida albicans detection rate | 6 months
  Candida albicans detection rate was defined as the percentage of patients in whose colonic mucosa candida albicans were identified.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sokol H, Leducq V, Aschard H, Pham HP, Jegou S, Landman C, Cohen D, Liguori G, Bourrier A, Nion-Larmurier I, Cosnes J, Seksik P, Langella P, Skurnik D, Richard ML, Beaugerie L. Fungal microbiota dysbiosis in IBD. Gut. 2017 Jun;66(6):1039-1048. doi: 10.1136/gutjnl-2015-310746. Epub 2016 Feb 3. PMID 26843508
- [Result] Mukhopadhya I, Hansen R, Meharg C, Thomson JM, Russell RK, Berry SH, El-Omar EM, Hold GL. The fungal microbiota of de-novo paediatric inflammatory bowel disease. Microbes Infect. 2015 Apr;17(4):304-10. doi: 10.1016/j.micinf.2014.12.001. Epub 2014 Dec 15. PMID 25522934
- [Result] Eriksson M, Johannssen T, von Smolinski D, Gruber AD, Seeberger PH, Lepenies B. The C-Type Lectin Receptor SIGNR3 Binds to Fungi Present in Commensal Microbiota and Influences Immune Regulation in Experimental Colitis. Front Immunol. 2013 Jul 16;4:196. doi: 10.3389/fimmu.2013.00196. eCollection 2013. PMID 23882266
- See also: PUBmed — http://www.ncbi.nlm.nih.gov/pubmed?term=fungal%20microbiota%20disbiosis%20in%20ibd&cmd=correctspelling
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=The+fungal+microbiota+of+de-novo+paediatric+inflammatory+bowel+disease